CLINICAL TRIAL: NCT06473116
Title: Epinephrine Versus Isoprenaline During Out-of-Hospital Cardiac Arrest With Asystole: A Randomized Clinical Trial
Brief Title: Epinephrine Versus Isoprenaline During Out-of-Hospital Cardiac Arrest With Asystole
Acronym: EPISO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Laura Sarkisian Jangaard, MD, PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPISOTrial
Record Dates: First submitted 2024-06-05; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Isoproterenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Isoprenaline
  Interventions: Drug: Isoprenaline Only Product
- Control group (Active Comparator): Epinephrine (adrenaline)
  Interventions: Drug: Isoprenaline Only Product

INTERVENTIONS:
Drug: Isoprenaline Only Product — Administration of intravenous isoprenaline of 600 mikrograms immediately after recognition of asystole in bystander-witnessed out-of-hospital cardiac arrest
  Other Names: isoproterenol

SUMMARY:
Background: During out-of-hospital cardiac arrest (OHCA), the patient presents with either a shockable or a non-shockable rhythm. Early cardiopulmonary resuscitation (CPR) and defibrillation of the shockable rhythm may increase chance of survival to more than 50%, however, if untreated, the heart rhythm will deteriorate to a non-shockable rhythm with dismal survival outcomes of 1-5%. Isoprenaline is a pro-arrhythmic drug used to treat bradycardia, and has a structural resemblance to epinephrine, which is the drug of choice during cardiac arrest with non-shockable rhythms.

Aims: To evaluate whether intravebous (IV) administration of isoprenaline increases the chance of return of spontaneous circulation (ROSC) to hospital arrival (main outcome) compared with IV epinephrine.

Study design: A randomized-controlled trial.

Setting: The study will be conducted in the Region of Southern Denmark, which has about 1.2 million inhabitants and an annual incidence of 1,200 OHCAs. The study will include bystander-witnessed patients with asystole at the arrival of the emergency medical services (EMS). Randomization will take place on arrival of the EMS, where the OHCA patients randomly will be assigned to receive an intravenous injection of isoprenaline (600 µg) or an intravenous injection of adrenaline (1 mg) in a 1:1 ratio. The study will include 1,178 OHCAs over a time period of about 3.5 years.

DETAILED DESCRIPTION:
Background: Out-of-hospital cardiac arrest (OHCA) is the leading cause of death in industrialized countries. During OHCA, the patient will present with either a non-shockable or a shockable rhythm. A shockable rhythm is treated by defibrillation, which means delivering an electrical shock through the heart to reestablish normal cardiac electric activity. If a shockable rhythm is defibrillated early, chances of survival can exceed 50%. However, if the shockable rhythm remains untreated, it will deteriorate into a non-shockable rhythm with dismal survival rates of 1-5%. Epinephrine increases the chance of return of spontaneous circulation (ROSC), however, there is increasing evidence that use of epinephrine is associated with severe neurological impairment in survivors. Isoprenaline is a pro-arrhythmic drug used to treat bradycardia. The drug has structural resemblance to epinephrine, however, it has no effect on alfa-adrenoceptors in the cerebral bloodflow and only stimulates beta-adrenoceptors. These pro-arrhythmic properties may induce cardiac electrical activity during OHCA with a non-shockable rhythm, converting it to a shockable rhythm treatable by defibrillation, while preserving microcirculatory cerebral blood flow.

Hypothesis: Injection of isoprenaline in bystander witnessed OHCAs with asystole increases the chance of ROSC at hospital arrival compared with the injection of epinephrine.

Population: According to the Danish Cardiac Arrest Registry, the annual incidence of OHCAs in the Region of Southern Denmark is about 1200, half of which are bystander witnessed. In the recent 2022 report, the incidence of non-shockable first rhythm among these was 1,044 out of 1,233 patients (85%), of which about 9 out of 10 had asystole. Therefore, an annual number of 450 bystander witnessed OHCAs with non-shockable rhythm could be eligible for study entry, however, despite eligibility, previous study have found that about 20-25% of patients are not enrolled in similar OHCA trials, and the expected annual number of enrollments will therefore be 360 OHCAs.

Settings: The study will take place in the Region of Southern Denmark. The Region has 42 EMS ambulance stations and 6 physician-manned vehicles with a median response time of about 8 minutes. The EMS ambulance has an emergency medical technician (EMT) and an EMT assistant, trained in analysing shockable/non-shockable rhythms and administering intravenous drugs according to the advanced life support algorithm.

Intervention: On EMS arrival, OHCA patients will be randomly assigned to receive an intravenous injection of isoprenaline or to receive an intravenous injection of adrenaline in a 1:1 ratio.

Study design: A randomized-controlled trial.

Main outcome: Main outcome is ROSC at hospital arrival. Secondary outcomes are conversion from non-shockable to shockable rhythm, 30-day survival with good neurological outcome (Cerebral Performance Category Scale of 1 or 2).

Power analysis: Thirty-day survival among OHCAs with non-shockable rhythm is reported at 1-5%. In a Danish study, the conversion of a non-shockable rhythm to a shockable rhythm increased the rate of ROSC at hospital arrival to 14.5% compared with 8.4% for sustained non-shockable rhythms. Thirty-day survival in the two groups were 4.2% versus 1.2%, respectively. According to this study, about 1 in 8 non-shockable rhythms converted to a shockable rhythm. Presuming that isoprenaline injection may double the conversion to shockable rhythm to 1 in 4 non-shockable rhythms, this would increased chance of ROSC at hospital arrival to approximately 13%. Therefore, assuming a conservative difference estimate of about 5% (estimate of 13% in the intervention group and 8% in the control group), this study will require a total sample size of 1178 patients with 589 OHCAs in each group (power value of 0.80 and significance level of 0.05) to evaluate the hypothesis. An inclusion time of approximately 3.5 years is therefore to be expected.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed out-of-hospital cardiac arrest
* Age 18 years or more
* Initial rhythm asystole at EMS arrival
* Advanced life support initiated or continued by EMS personnel

Exclusion Criteria:

* Cardiac arrest caused by blunt trauma, penetrating trauma, or burn injury suspected to be the cause of the cardiac arrest
* Cardiac arrest caused by drowning, hanging, strangulation, and foreign body airway obstruction
* IV epinephrine already administered prior to EMS arrival
* Prior enrollment in the trial
* Known or apparent pregnancy
* Cardiac arrest at nursing homes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1178 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Return of Spontaneous Circulation (ROSC) at hospital arrival | Up to 2 hours
  Arrival to hospital admission

SECONDARY OUTCOMES:
Rate of conversions from asystole to shockable rhythm | Up to 1 hour
  The conversion from asystole to either pulseless ventricular tachycardia or ventricular fibrillation during cardiac arrest resuscitation
Number of participants with favorable neurological outcome at hospital discharge | Median hospital stay is about 24 days after out-of-hospital cardiac arrest
  The modified Rankin Scale (mRS) is ranked from 0 to 6 and defined the following way: A score of 0) represents no symptoms; 1) no significant disability; 2) slight disability; 3) moderate disability; 4) moderately severe disability; 5) severe disability and 6) death. Favorable neurological outcome is defined as mRS score of 0-3.
TNumber of participants alive after 30 days | At 30 days
  Survival at 30 days after the out-of-hospital cardiac arrest
Number of participants who gain sustained return of spontaneous circulation | 20-50 minutes
  The patient achieved sustained return of spontaneous circulation (ROSC), defined as ROSC of at least 20 minutes after the cardiac arrest. ROSC is defined as the resumption of a sustained heart rhythm that perfuses the body after cardiac arrest.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Department of Cardiology, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Six months after the publication of the last results, all de-identified individual patient data will be made available for data sharing, and there will be no predetermined end date for the data sharing. Data will be completely anonymized according to Danish law. The main protocol, data dictionary for the REDCap database and the statistical analyses will also be made available. Interested parties with appropriate approval and methodologically sound proposals will be able to request the trial data by contacting the principal investigator and considered for data sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after the publication of the last results.
Access Criteria: Appropriate approval of the study and methodologically sound proposals will be able to request the trial data by contacting the principal investigator and considered for data sharing.